CLINICAL TRIAL: NCT06079320
Title: AN INTERVENTIONAL PHASE 2/3, ADAPTIVE, MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND STUDY TO INVESTIGATE EFFICACY AND SAFETY OF ORAL SISUNATOVIR COMPARED WITH PLACEBO IN NON-HOSPITALIZED SYMPTOMATIC ADULTS WITH RESPIRATORY SYNCYTIAL VIRUS INFECTION WHO ARE AT RISK OF PROGRESSION TO SEVERE ILLNESS
Brief Title: A Study to Learn About the Study Medicine Sisunatovir in Adults With Respiratory Syncytial Virus (RSV) Infection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study discontinued due to business reasons. There were no safety concerns in the decision to stop study and no changes to sponsor's assessment of the risk-benefit profile for participants who received sisunatovir in the study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C5241007; 2023-505922-32-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — sisunatovir

STUDY DESIGN:
Intervention Model Description: This is a Phase 2/ Phase 3, superiority, adaptive, two parallel-arm, randomized, multi-center, placebo-controlled, double-blind study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be assigned to receive study intervention according to the assigned treatment group from the randomization scheme. Investigators will remain blinded to each participant's assigned study intervention until all participants complete treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sisunatovir (Experimental)
  Interventions: Drug: Sisunatovir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sisunatovir — Participants will receive tablets from Day 1 to Day 5
  Arms: Sisunatovir
Drug: Placebo — Participants will receive matching placebo tablets from Day 1 to Day 5
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the safety and effects of sisunatovir. Sisunatovir is studied for the possible treatment of Respiratory Syncytial Virus (RSV). RSV is a virus that causes lung infections with cold-like symptoms, but it can cause severe illness in some people. Sisunatovir is studied in adults:

* who are not admitted to the hospital and
* who have high chances of having a severe illness from RSV infection.

This study is seeking participants who:

* Are confirmed to have RSV.
* Have symptoms of a lung infection.
* Are 18 years of age or older.
* Have one or more of the following which increases the chances of RSV illness:
* A long-term lung disease.
* heart failure.
* a condition that weakens the immune system.
* Are 65 years of age or older and do not have any of the conditions above

Half of the participants in this study will receive sisunatovir. The other half will receive a placebo for 5 days. Placebo looks same like the study medicine but does not have any medication. Both sisunatovir and placebo will be taken by mouth. The study will compare the experiences of people receiving sisunatovir to those of the people who do not. This will help decide if sisunatovir is safe and effective.

Participants will attend about 8-10 study visits over 5 weeks. During this time, they will have:

* visits at the study clinic,
* blood work,
* swabs of the nose,
* questionnaires,
* a follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older at screening.
* Diagnosis of RSV infection collected within 5 days prior to randomization.
* New onset or worsening (if present chronically) of at least one of the following signs and/or symptoms consistent with a viral acute respiratory infection (ARI), within 5 days prior to randomization: nasal congestion, nasal discharge, sore throat, cough, sputum production, shortness of breath, or wheezing.
* Has at least 1 of the following characteristics or underlying medical conditions: a) 65 years of age or older b) Chronic lung disease, c) Heart failure, d) Immunosuppressive disease/condition or immune-weakening medications

Exclusion Criteria:

* Any medical or psychiatric condition that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study or interfere with the evaluation of response to the study intervention.
* Diagnosis of viral respiratory infections other than RSV including influenza and SARS-CoV-2
* Current need for hospitalization or anticipated need for hospitalization for any reason to provide inpatient/acute care within 24 hours after randomization
* Any clinically significant ECG abnormality in the pre-dose ECG that, per investigator judgement, may affect participant safety
* Has hypersensitivity to or other contraindication to any of the components of the study interventions, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (14):
  - National Institute of Clinical Research, Garden Grove, California
  - National Institute of Clinical Research, Westminster, California
  - De La Cruz Research Center, LLC, Miami, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Adult Medicine of Lake County, Mt. Dora, Florida
  - Accellacare - DuPage, Oak Lawn, Illinois
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - DM Clinical Research - AOM, Brooklyn, New York
  - CHEAR Center LLC, The Bronx, New York
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Zenos Clinical Research, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Salma Mazhar, MD PA, Mesquite, Texas
  - SMS Clinical Research, Mesquite, Texas
- Shanghai Minhang District Central Hospital, Shanghai, China
- Maharaja Agrasen Superspeciality Hospital, Jaipur, Rajasthan, India
- Japan (3):
  - Koukankai Koukan Clinic, Kawasaki-Shi, Kanagawa
  - National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto
  - Nanbu Tokushukai Hospital, Shimajiri, Okinawa

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 participants were enrolled at 16 centers in the United States, China, Japan and India.
Groups:
- Sisunatovir: Participants received oral doses of sisunatovir from Day 1 to Day 5.
- Placebo: Participants received oral doses of placebo from Day 1 to Day 5.
Period: Treatment Phase
Arm/Group | Sisunatovir | Placebo
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Follow up Phase
Arm/Group | Sisunatovir | Placebo
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sisunatovir | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (10.96) | 60.8 (9.13) | 62.3 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Syncytial Virus (RSV) Related Hospitalization or Death From Any Cause Through Day 28
Description: RSV related hospitalization included a specialized acute medical care unit within an assisted living facility or nursing home.
Time Frame: From Day 1 (start of study intervention) up to Day 28
Population: Modified Intent-to-Treat-Infected (mITT-infected) population included all participants randomly assigned to study intervention, who took at least 1 dose of study intervention, and who had confirmed RSV infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With RSV-Related Visits (Urgent Care/ Emergency Department (ED)/Hospital) or Death From Any Cause Through Day 28
Description: Participants with RSV related visits in a hospital/urgent care or ED requiring no minimum duration of hospitalization were reported in this outcome measure. Investigators determined if a medical visit was related to RSV. RSV-related medical visits were those attendances that would not otherwise occur in the absence of the RSV infection. These may have included: deterioration or decompensation of the lung function that required supplemental oxygen; development of secondary respiratory tract infections that required antibiotic treatment; management of severe symptoms associated with RSV such as fever; worsening or decompensation of cardiac or renal function in participants with underlying cardiac or renal disease.
Time Frame: From Day 1 (start of study intervention) up to Day 28
Population: mITT-infected population included all participants randomly assigned to study intervention, who took at least 1 dose of study intervention, and who had confirmed RSV infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Progression of Lower Respiratory Tract Infection (LRTI) Through Day 10
Description: Progression of LRTI was defined as development of LRTI or transition from non-severe LRTI-RSV at randomization to severe LRTI-RSV at any time up to and including Day 10. LRTI was defined as: >= 2 lower respiratory signs or symptoms for at least 24 hours including at least 1 lower respiratory sign; or 3 lower respiratory symptoms for at least 24 hours. Lower respiratory symptoms included following: new or increased sputum, new or increased cough, new or increased dyspnea (shortness of breath). Lower respiratory signs included: new or increased wheezing, new or increased crackles/ronchi based on chest auscultation, respiratory rate >= 20 respirations/minute, low or decreased oxygen saturation (O2 less than (<) 95 percent (%) or <= 90% if pre-season baseline is < 95%), need for new or increased oxygen supplementation.
Time Frame: From randomization on Day 1 up to Day 10
Population: mITT-infected population included all participants randomly assigned to study intervention, who took at least 1 dose of study intervention, and who had confirmed RSV infection. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Development of LRTI Through Day 10
Description: Development of LRTI was defined as transitioning from not having LRTI at randomization but having nsLRTI-RSV or sLRTI-RSV at any time up to and including Day 10. LRTI was defined as: >= 2 lower respiratory signs or symptoms for at least 24 hours including at least 1 lower respiratory sign; or 3 lower respiratory symptoms for at least 24 hours. Lower respiratory symptoms included following: new or increased sputum, new or increased cough, new or increased dyspnea (shortness of breath). Lower respiratory signs included: new or increased wheezing, new or increased crackles/ronchi based on chest auscultation, respiratory rate >= 20 respirations/minute, low or decreased oxygen saturation (O2 < 95 % or <= 90% if pre-season baseline is < 95%), need for new or increased oxygen supplementation.
Time Frame: From randomization on Day 1 up to Day 10
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Resolution of LRTI at Day 15
Description: Resolution of LRTI was defined as transition from RSV-related non-severe LRTI (nsLRTI-RSV) or RSV-related severe LRTI (sLRTI-RSV) at randomization to not having nsLRTI and sLRTI-RSV. LRTI was defined as: >= 2 lower respiratory signs or symptoms for at least 24 hours including at least 1 lower respiratory sign; or 3 lower respiratory symptoms for at least 24 hours. Lower respiratory symptoms included following: new or increased sputum, new or increased cough, new or increased dyspnea (shortness of breath). Lower respiratory signs included: new or increased wheezing, new or increased crackles/ronchi based on chest auscultation, respiratory rate >= 20 respirations/minute, low or decreased oxygen saturation (O2 < 95 % or <= 90% if pre-season baseline is < 95%), need for new or increased oxygen supplementation.
Time Frame: Day 15
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 3 | 3
Participants | 1 | 1

6. Secondary Outcome: Mean Number of Hospital Free Days Through Day 28
Time Frame: From Day 1 (start of study intervention) up to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Days | 28.0 (0.00) | 28.0 (0.00)

7. Secondary Outcome: Number of Participants With Progression of LRTI Through Days 3, 5, 15 and 28
Description: Progression of LRTI was defined as development of LRTI or transition from non severe LRTI-RSV at randomization to severe LRTI-RSV at any time up to and including Days 3, 5, 15 and 28. LRTI was defined as: >= 2 lower respiratory signs or symptoms for at least 24 hours including at least 1 lower respiratory sign; or 3 lower respiratory symptoms for at least 24 hours. Lower respiratory symptoms included following: new or increased sputum, new or increased cough, new or increased dyspnea (shortness of breath). Lower respiratory signs included: new or increased wheezing, new or increased crackles/ronchi based on chest auscultation, respiratory rate >= 20 respirations/minute, low or decreased oxygen saturation (O2 < 95 % or <= 90% if pre-season baseline is < 95%), need for new or increased oxygen supplementation.
Time Frame: From randomization on Day 1 up to Days 3, 5, 15 and 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 3
Participants
  Day 3 | 0 | 0
  Day 5 | 0 | 0
  Day 15 | 0 | 0
  Day 28 | 0 | 0

8. Secondary Outcome: Number of Participants With Development of LRTI Through Days 3, 5, 15 and 28
Description: Development of LRTI was defined as transitioning from not having LRTI at randomization but having nsLRTI-RSV or sLRTI-RSV at any time up to and including Days 3, 5, 15 and 28. LRTI was defined as: >= 2 lower respiratory signs or symptoms for at least 24 hours including at least 1 lower respiratory sign; or 3 lower respiratory symptoms for at least 24 hours. Lower respiratory symptoms included following: new or increased sputum, new or increased cough, new or increased dyspnea (shortness of breath). Lower respiratory signs included: new or increased wheezing, new or increased crackles/ronchi based on chest auscultation, respiratory rate >= 20 respirations/minute, low or decreased oxygen saturation (O2 < 95 % or <= 90% if pre-season baseline is < 95%), need for new or increased oxygen supplementation.
Time Frame: From randomization on Day 1 up to Days 3, 5, 15 and 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 1 | 2
Participants
  Day 3 | 0 | 0
  Day 5 | 0 | 0
  Day 15 | 0 | 0
  Day 28 | 0 | 0

9. Secondary Outcome: Number of Participants With Resolution of LRTI at Days 3, 5, 10 and 28
Description: Resolution of LRTI was defined as transition from nsLRTI-RSV or sLRTI-RSV at randomization to not having nsLRTI and sLRTI-RSV. LRTI was defined as >= 2 lower respiratory signs or symptoms for at least 24 hours including at least 1 lower respiratory sign; or 3 lower respiratory symptoms for at least 24 hours. Lower respiratory symptoms included following: new or increased sputum, new or increased cough, new or increased dyspnea (shortness of breath). Lower respiratory signs included: new or increased wheezing, new or increased crackles/ronchi based on chest auscultation, respiratory rate >= 20 respirations/minute, low or decreased oxygen saturation (O2 < 95% or <= 90% if pre-season baseline is < 95%), need for new or increased oxygen supplementation.
Time Frame: At Days 3, 5, 10 and 28
Population: mITT-infected population included all participants randomly assigned to study intervention, who took at least 1 dose of study intervention, and who had confirmed RSV infection. Here, "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 3 | 3
Participants
  Day 3 | 1 | 1
  Day 5 | 1 | 1
  Day 10 | 1 | 1
  Day 28 | 2 | 3

10. Secondary Outcome: Number of Participants With Improvement of LRTI at Days 3, 5, 10, 15 and 28
Description: Improvement in LRTI status was defined as LRTI resolution or transition from sLRTI-RSV at randomization to nsLRTI-RSV. LRTI was defined as: >= 2 lower respiratory signs or symptoms for at least 24 hours including at least 1 lower respiratory sign; or 3 lower respiratory symptoms for at least 24 hours. Lower respiratory symptoms included following: new or increased sputum, new or increased cough, new or increased dyspnea (shortness of breath). Lower respiratory signs included: new or increased wheezing, new or increased crackles/ronchi based on chest auscultation, respiratory rate >= 20 respirations/minute, low or decreased oxygen saturation (O2 < 95 % or <= 90% if pre-season baseline is < 95%), need for new or increased oxygen supplementation.
Time Frame: At Days 3, 5, 10, 15 and 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 3 | 3
Participants
  Day 3 | 1 | 2
  Day 5 | 1 | 2
  Day 10 | 1 | 2
  Day 15 | 1 | 3
  Day 28 | 2 | 3

11. Secondary Outcome: Mean Number of RSV Related Days in Hospital Through Day 28
Description: as for outcome 1
Time Frame: From Day 1 (start of study intervention) up to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Days | 0 (0) | 0 (0)

12. Secondary Outcome: Mean Number of RSV Related Days in Intensive Care Unit (ICU) Through Day 28
Time Frame: From Day 1 (start of study intervention) up to Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Days | 0 (0) | 0 (0)

13. Secondary Outcome: Number of Participants With a Clinical Response of Improvement or Resolution at Days 5, 10, 15, and 28
Description: Improvement was defined as no new acute respiratory infection (ARI) signs or symptoms, and no worsening of existing signs or symptoms compared to the Day 1 visit. At least one sign or symptom (but not all) present at Day 1 was absent, improved or returned to pre-infection status. Resolution was defined as all ARI signs or symptoms were absent or returned to pre-infection status. Clinical response was evaluated by the investigator.
Time Frame: At Days 5, 10, 15, and 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Participants
  Day 5 | 3 | 5
  Day 10 | 4 | 5
  Day 15 | 3 | 5
  Day 28 | 3 | 5

14. Secondary Outcome: Number of Participants With Undetectable RSV Viral Load at Days 3, 5, 10, 15 and 28
Description: Undetectable RSV viral load at a visit was defined as a central PCR laboratory result of target not detected (TND).
Time Frame: At Days 3, 5, 10, 15, and 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Participants
  Day 3 | 0 | 0
  Day 5 | 0 | 1
  Day 10 | 1 | 2
  Day 15 | 4 | 5
  Day 28 | 4 | 5

15. Secondary Outcome: Change From Baseline in Log10 Transformed Total RSV Viral Load at Days 3, 5, 10, 15 and 28
Description: Undetectable viral load was considered to be 0 copies/mL for this analysis.
Time Frame: Baseline (within 1 hour post start of study intervention on Day 1) and Days 3, 5, 10, 15, and 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 4 | 5
Log10 copies/mL
  Day 3 | -1.453 (1.2107) | -1.184 (1.2960)
  Day 5 | -1.788 (2.0327) | -1.626 (1.6493)
  Day 10 | -4.445 (1.5779) | -2.784 (1.8207)
  Day 15 | -6.110 (2.6486) | -4.900 (1.7815)
  Day 28 | -6.110 (2.6486) | -4.900 (1.7815)

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Through Day 35
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An adverse event was considered a TEAE if the event started on or after the study intervention start date (Day 1).
Time Frame: From Day 1 of study intervention up to 28-30 days after last dose of study drug (up to Day 35)
Population: Safety analysis set (SAS) included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 1 | 4

17. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAE) Through Day 35
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the criteria listed below: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic and other important medical event.
Time Frame: From Day 1 of study intervention up to 28-30 days after last dose of study drug (up to Day 35)
Population: SAS included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

18. Secondary Outcome: Plasma Concentrations of Sisunatovir at Days 3 and 5
Time Frame: Anytime between 3 to 8 hours post dose on Day 3, and pre-dose on Day 5
Population: Pharmacokinetic (PK) concentration analysis set included all participants who received at least 1 dose of sisunatovir and in whom at least 1 concentration value was reported. Here, "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Sisunatovir
Number analyzed (Participants) | 7
Nanogram per milliliter
  Day 3 | 98.26 (141.41)
  Day 5: number analyzed (Participants) | 5
  Day 5 | 173.1 (231.83)

ADVERSE EVENTS:
Time Frame: From Day 1 of study intervention up to 28-30 days after last dose of study drug (up to Day 35)
Description: SAS included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | Sisunatovir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sisunatovir (N=8) | Placebo (N=8)
Constipation (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
A limitation of these results was the early study termination. Due to the small sample size, the study was no longer powered to establish the efficacy for the primary and key secondary efficacy endpoints for sisunatovir compared to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT06079320/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT06079320/SAP_001.pdf